CLINICAL TRIAL: NCT02630758
Title: Mindfulness-Based Yoga Intervention for Women With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1203P11124
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Depressive Symptoms
Keywords: depression; yoga; mindfulness
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based Yoga (Experimental): Participants in the 12-week mindfulness-based yoga condition were guided by a gentle yoga DVD that included postures (asanas), pranayama (breathing exercises), and relaxation (meditation). Participants were asked to complete 60-75 minutes of the DVD twice per week and were encouraged to do more if they were interested.
  Following the initial baseline assessment and randomization telephone interview, participants in the yoga group completed weekly 15-minute telephone sessions for the first month and bi-weekly telephone sessions for the second and third for a total of eight sessions over the 12 weeks. The mindfulness telephone sessions were modified from the Mindfulness-Based Stress Reduction.
  Interventions: Behavioral: Mindfulness-based Yoga
- Walking Control Group (Active Comparator): The 12-week walking control condition included twice-weekly home practice with a 65-minute walking DVD (Sansone, 2008) and eight telephone sessions with the telephone counselor.
  Participants were asked to complete 60 minutes of the DVD (or other walking) twice weekly and encouraged to do more if they were interested.
  Participants received telephone sessions on the same schedule as the yoga condition. The education sessions covered a variety of health and wellness related topics.
  Interventions: Behavioral: Walking Control Condition

INTERVENTIONS:
Behavioral: Mindfulness-based Yoga — See study arm description.
  Arms: Mindfulness-based Yoga
Behavioral: Walking Control Condition — See study arm description.
  Arms: Walking Control Group

SUMMARY:
The purpose of this study was to examine the efficacy of a 12-week mindfulness-based yoga intervention on depressive symptoms and rumination among depressed women.

DETAILED DESCRIPTION:
This study was a prospective, randomized controlled intervention pilot study conducted in a metropolitan city in the upper Midwest of the United States. Forty women who met the criteria for depression based on the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders IV (SCID-I; First, Spitzer, Gibbon, & Williams, 1997)were randomized to an experimental mindfulness-based yoga condition (n=20) or a walking control condition (n=20). Both programs were home-based motivational sessions delivered over the telephone and lasted 12 weeks. Assessments were conducted at baseline, three months (i.e., post-intervention), one-month follow-up (i.e., one month after the intervention ended). Participants were instructed to continue their usual depression care. The primary dependent variable was depressive symptoms based on the Beck Depression Inventory (BDI). The secondary dependent variable was rumination scores on the Ruminative Responses Scale (RRS). This protocol was approved by the University of Minnesota's Institutional Review Board (IRB). Participants completed informed consent forms sent through the mail; consent to participate in physical activity was also obtained from the participant's healthcare provider. Recruitment for this trial occurred from February, 2013 to January, 2014 and follow-up assessments were completed by May, 2014.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* a personal history of depression (i.e., ever being told by a healthcare provider that they had depression or given an antidepressant for depression)
* able to read and write in the English language
* able to commit to two sessions (yoga or walking) per week for 12 weeks
* demonstrate a willingness to be randomly assigned to either of the study arms
* be yoga naïve, defined as not taking more than four yoga classes in the past two years and not more than one class in the past month.

Exclusion Criteria:

* individuals with a history of bipolar disorder or schizophrenia and/or who had been hospitalized for a psychiatric disorder within six months prior to the eligibility screening
* individuals not providing signed informed consent
* individuals reporting any other health problems that would interfere with regular yoga practice or walking sessions
* individuals who engaged in more than 90 minutes of moderate intensity physical activity per week during the month prior to the eligibility screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory | 3 months
  Change from Baseline Depression at 3 months

SECONDARY OUTCOMES:
Ruminative Responses Scale | 3 months
  Change from Baseline Rumination at 3 months
Five Facet Mindfulness Questionnaire | 3 months
  Change from Baseline Mindfulness at 3 months
Perceived Stress Scale | 3 months
  Change from Perceived Stress at 3 months
Pittsburgh Sleep Scale | 3 months
  Change from Baseline Sleep at 3 months
Quality of Life Enjoyment and Satisfaction Questionnaire- Short Form | 3 months
  Change from Baseline Quality of LIfe Enjoyment and Satisfaction at 3 months

OTHER OUTCOMES:
Body Mass Index | 3 months
  Change from Baseline Body Mass Index at 3 months
7-Day Physical Activity Recall | 3 months
  Change from Baseline Physical Activity at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Lewis, PHD, L.P., Study Chair — University of Minnesota

IPD SHARING:
Plan to Share IPD: No